CLINICAL TRIAL: NCT06748612
Title: Immunogenicity of Different Primary Immunization Schedules with Inactivated Poliovirus Vaccine (IPV) Plus Pentavalent Vaccine (DTwP-HBV-Hib) or with Hexavalent Vaccine (DTwP-HBV-Hib-IPV)
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: PR-24093
Record Dates: First submitted 2024-11-25; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-10

CONDITIONS: Polio
MeSH Terms: conditions — Poliomyelitis | interventions — Vaccines, Combined; Poliovirus Vaccine, Inactivated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm A (Experimental): Arm A will receive wP-Penta at 6,10,14 weeks of age and 2 doses of IPV at 14 weeks and 9 months.
  Interventions: Biological: Pentavalent vaccine; Biological: Inactivated poliovirus vaccine (IPV)
- Arm B (Experimental): Arm B will receive wP-Hexa at 6,10,14 weeks of age
  Interventions: Biological: Hexavalent vaccine
- Arm C (Experimental): Arm C will receive wP-Hexa at 2,4,6 months of age.
  Interventions: Biological: Hexavalent vaccine
- Control Arm (Active Comparator): Control group will receive EPI schedule of routine immunization: fIPV @ 6, 14 wk, bOPV @ 6, 10, 14 wk , wP-Penta @ 6, 10, 14 wk
  Interventions: Biological: Pentavalent vaccine; Biological: Bivalent oral polio vaccine (bOPV); Biological: Fractional IPV( fIPV)

INTERVENTIONS:
Biological: Pentavalent vaccine — Whole-cell pertussis pentavalent vaccine (wP-Penta): Each 0.5 ml dose contains diphtheria toxoid, Tetanus toxoid, whole cell pertussis, Hepatitis B surface antigen, Haemophilus influenzae type b conjugate
  Arms: Arm A; Control Arm
Biological: Hexavalent vaccine — Whole-cell pertussis hexavalent vaccine (wP-Hexa): Each 0.5 ml dose contains diphtheria toxoid, Tetanus toxoid, whole cell pertussis, Hepatitis B surface antigen, Haemophilus influenzae type b conjugate, and inactivated polioviruses to all three poliovirus types: type 1 , 2 and 3
  Arms: Arm B; Arm C
Biological: Inactivated poliovirus vaccine (IPV) — one dose of IPV (0.5 mL) contains inactivated polioviruses to all three poliovirus types: type 1, 2 and 3
  Arms: Arm A
Biological: Bivalent oral polio vaccine (bOPV) — Contain two poliovirus types: type 1 and 3
  Arms: Control Arm
Biological: Fractional IPV( fIPV) — The dose of fIPV is 0.1 mL or 1/5th of a full dose
  Arms: Control Arm

SUMMARY:
The goal of this study is to provide information on immunogenicity at short and medium term for hexavalent with different schedules, which will be useful for the global polio program and countries, including Bangladesh.

Primary objectives are

1. To compare the proportion of participants who seroconvert to all poliovirus serotypes four weeks after a primary immunization series.
2. To compare the proportion of participants seropositive against all poliovirus serotypes at 18 months of age.

This is an open-label randomized clinical trial. Participants will be enrolled and randomized at 6 weeks of age to one of three arms. Target enrolment is 330 infants per arm and 200 controls; 990 in the main study and ~ 800 in the sub-study.

A total of 4-5 blood samples will be collected from each infant before and after the primary vaccination series, and at 18 months of age, to assess systemic immune response to different antigens.

Outcome measures/variables:

Neutralizing antibody titers in serum will be quantified for poliovirus types 1, 2, and 3 using a microneutralization test; for diphtheria toxoid, tetanus toxoid, and pertussis toxin using a Multiplex bead assay; and for antibodies to hepatitis B surface antigen (anti-HBs) using serologic assay. The presence of poliovirus types 1 and 3 in oropharyngeal swabs and stools following the bOPV challenge will be tested using a real-time reverse transcription PCR (rRT-PCR) assay.

DETAILED DESCRIPTION:
After eradicating wild poliovirus, the inactivated poliovirus vaccine (IPV) which contains killed poliovirus will replace the oral poliovirus vaccine (OPV) containing attenuated strains in routine immunization to avoid paralysis caused by vaccine-derived polioviruses. However, although IPV is safe and induces high levels of serum antibodies that provide long-term protection against polio, it is less effective in providing mucosal immunity required to prevent person-to-person transmission. Inclusion of IPV in routine immunization schedules in many low-income countries also requires additional injections per visit and delaying of doses to avoid interference of maternally-derived antibody titers.

Introduction of recently licensed hexavalent vaccines containing whole-cell Pertussis, Diphtheria toxoid, Tetanus toxoid, Hepatitis B, Haemophilus influenza type B and IPV (wP-Hexa), could reduce the number of vaccine injections per visit, potentially increasing coverage for polio vaccination in low and middle-income countries currently using pentavalent plus stand-alone IPV. But there is limited data on immunogenicity for long-term protection against polio and other antigens with wP-Hexa administered in early short vaccination schedules (i.e. 6-10-14 weeks) without boosters.

Investigators need additional research on safety and immunogenicity across different schedules of IPV containing wP-Hexa, to assist countries in making informed decisions for vaccine introduction. Investigators also need more information on oropharyngeal mucosal immunity induced by IPV alone to assess its effectiveness in preventing poliovirus transmission after importations in low, middle-income countries.

Primary Objectives:

1. To compare the proportion of participants who seroconvert to all poliovirus serotypes four weeks after a primary immunization series.
2. To compare the proportion of participants seropositive against all poliovirus serotypes at 18 months of age.

Secondary objectives:

1. To compare antibody titers for all polio serotypes at 18 months of age among study arms
2. To assess seroprotection/vaccine response for non-polio antigens contained in wP-Hexa or wP-Penta one month after a 3-dose vaccination series.
3. To assess seroprotection/antibody levels for non-polio antigens at 18 months of age following the primary series.
4. To assess solicited and unsolicited adverse effects.
5. Sub-study (Arms A, B and control group only): To compare the proportion of infants shedding type 1 and 3 poliovirus in oropharynx and stools following a challenge with bivalent oral poliovirus vaccine (bOPV).

The study will be an open label, phase IV, randomized, inequality, controlled trial.The study will be carried out in Dakshinkhan and Uttarkhan area of Dhaka North City Corporation (DNCC).Eligible infants will be identified through active surveillance of new births in the community and parents will be requested to participate through home visits by local field workers. Participants will be enrolled at 6 weeks of age, randomly assigned to one of three study arms, and followed up to 18 months of age.

Following parental informed consent, healthy infants from Dhaka, Bangladesh, will be randomized to one of 3 primary immunization schedules A, B, or C at 6 weeks of age:

* Arm A will receive wP-Penta at 6,10,14 weeks of age and 2 doses of IPV at 14 weeks and 9 months.
* Arm B will receive wP-Hexa at 6,10,14 weeks of age
* Arm C will receive wP-Hexa at 2,4,6 months of age. All participants will have 4-6 visits to the study clinic until 18 months of age. During each visit, the study staff will examine infants, obtain vaccination history and administer study vaccines. Blood collection will be done before and after the 3-dose series, at 10 months (for some antigens) and at 18 months of age.

In a subset of participants (those in study arms A and B), the bOPV dose administered to catch-up with the Bangladeshi essential immunization schedule will be used as a challenge dose to assess mucosal immunity induced by IPV. In addition, as a control arm, the study staff will enroll 200 children aged 18 months, who had received polio vaccination through routine immunization services verified by immunization card (bOPV at 6, 10 and 14 weeks; fIPV at 6 and 14 weeks).

All Study participants and controls will have a blood sample collected at 18 months, followed by a dose of bOPV (challenge dose) at the same visit. Then, participants in Arms A and B, and Controls, will attend the clinic 3 and 7 days after the challenge bOPV dose for an oropharyngeal swab. In addition, field workers will provide stool carriers with ice packs, a stool collection kit and instructions for parents to collect a stool sample from the baby and bring it to the clinic on day 7.

Outcome measures/variables:

Neutralizing antibody titers in serum will be quantified for poliovirus types 1, 2, and 3 using a microneutralization test; for diphtheria toxoid, tetanus toxoid, and pertussis toxin using a Multiplex bead assay; and for antibodies to hepatitis B surface antigen (anti-HBs) using serologic assay. The presence of poliovirus types 1 and 3 in oropharyngeal swabs and stools following the bOPV challenge will be tested using a real-time reverse transcription PCR (rRT-PCR) assay.

For assessing immunity to polio following the primary vaccination series, seroconversion will be defined as seronegative participants (<1:8 titers) becoming seropositive (≥1:8 titers) or seropositive participants with ≥ 4- fold increase in titers (adjusted for the expected decline of maternal antibodies) between pre-vaccination and four weeks after the third vaccine dose. Thresholds for seroprotection for other antigens will be: ≥0.1 IU for anti-diphtheria toxoid and anti-tetanus toxoid, ≥4-fold increase from baseline for pertussis toxin (and filamentous hemoglobin) and ≥ 10 mIU/mL for anti-HBs.

Solicited local and systemic reactions will be recorded 30 minutes and 48-72 hours after each vaccine dose; unsolicited adverse events will be collected throughout the study up to 18 months of age.

ELIGIBILITY:
A. Assessment of seroprotection and safety of wP-Hexa with primary immunization schedules.

Inclusion Criteria:

1. Healthy infants 6 weeks of age (range: 42-48 days).
2. Parents that consent for participation in the full length of the study.
3. Parents that can understand and comply with planned study procedures.

Exclusion Criteria:

1. Parents and infants are unable to participate in the full length of the study (e.g., plan to move away from the study area during the study period).
2. A diagnosis or suspicion of immunodeficiency disorder either in the infant or in an immediate family member.
3. A diagnosis or suspicion of bleeding disorder that would contraindicate administration of IPV, wP Penta or wP-Hexa, or collection of blood by venepuncture.
4. Acute diarrhoea, infection, or illness at the time of first study vaccination that would require infant's admission to a hospital.
5. Acute vomiting and intolerance to liquids within 24 hours before the first study vaccination.
6. Any encephalopathy of unknown origin occurring within 7 days following previous vaccination with any pertussis containing vaccine.
7. Uncontrolled neurologic disorder or uncontrolled epilepsy (Pertussis vaccine should not be administered to individuals with these conditions until the treatment regimen has been established and the condition has stabilized).
8. Evidence of a chronic medical condition identified by a study medical officer during physical exam.
9. Receipt of any polio vaccine (OPV or IPV) before enrolment based upon documentation or parental recall.
10. Known allergy/sensitivity or reaction to polio, pertussis, tetanus, diphtheria, hepatitis B, Hib vaccines or its contents.
11. Infants from multiple births. This exclusion is done because the non-participant infant will likely receive OPV through routine immunization and may transmit vaccine poliovirus to the enrolled infant.
12. Infants from premature births (<37 weeks of gestation).

B. Mucosal immunity against poliovirus sub-study :

Inclusion criteria

* Participants:

  * Participants in study arms A and B who complete study procedures up to 18 months and whose parents do not request discontinuation
* Controls:

  * Children aged 18 months who have received polio vaccination through routine immunization services verified by immunization card (bOPV at 6, 10 and 14 weeks; fIPV at 6 and 14 weeks)

Exclusion criteria

1. Parents and infants are unable to participate in the full length of the study (e.g., plan to move away from the study area during the study period).
2. A diagnosis or suspicion of immunodeficiency disorder either in the infant or in an immediate family member.
3. A diagnosis or suspicion of bleeding disorder that would contraindicate administration of bOPV or collection of blood by venepuncture.
4. Acute diarrhoea, infection, or illness at the time of enrolment (18 months of age) that would require infant's admission to a hospital.
5. Febrile disease that contraindicates administration of pentavalent vaccine (even if hospitalization is not required).
6. Acute vomiting and intolerance to liquids within 24 hours before the enrolment visit (18 months of age).
7. Known allergy/sensitivity or reaction to oral polio vaccines or its contents.
8. Received any polio vaccines outside of the routine immunization schedule.
9. Household members have received OPV within 1-2 months prior to enrolment.

Ages: 42 Days to 48 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1190 (Estimated)
Dates: Start 2025-01-28 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with seroconversion to all poliovirus serotypes four weeks after a primary immunization series with two doses of IPV or three doses of wP-Hexa | Arm A: 14 weeks and 10 months , Arm B: 6 and 18 weeks , Arm C: 2 and 7 months
  Seroconversion will be defined as seronegative participants (<1:8 titers) becoming seropositive (≥1:8) or seropositive participants with ≥ 4-fold increase in titers between pre vaccination and four weeks after the third vaccine dose (adjusted for the expected decline of maternal antibodies). For assessing immunity to polio, seropositivity is defined as reciprocal polio neutralizing antibody titers of at least 1:8. Baseline maternally-related antibody titers will be determined in the pre-vaccination sample and estimated maternal antibody level after the vaccination series will be calculated assuming an exponential decline with a half-life of 28 days
Proportion of participants seropositive to all polio types at 18 months of age (9-14 months after the last dose of IPV for each schedule). | 18 months for all study arms
  Seroconversion will be defined as seronegative participants (<1:8 titers) becoming seropositive (≥1:8) or seropositive participants with ≥ 4-fold increase in titers between pre vaccination and four weeks after the third vaccine dose (adjusted for the expected decline of maternal antibodies). For assessing immunity to polio, seropositivity is defined as reciprocal polio neutralizing antibody titers of at least 1:8. Baseline maternally-related antibody titers will be determined in the pre-vaccination sample and estimated maternal antibody level after the vaccination series will be calculated assuming an exponential decline with a half-life of 28 days

SECONDARY OUTCOMES:
Proportion of participants with seroprotection/vaccine response for non-polio antigens (Pertussis, Hepatitis B, Diphtheria, Tetanus) contained in wP-Hexa or wP-Penta four weeks after the last dose of wP-Hexa or wP-Penta | 6 and 18 weeks for A and B; 2 and 7 months for C
  Thresholds for seroprotection for other antigens will be: ≥0.1 IU for anti-diphtheria toxoid and anti-tetanus toxoid, ≥4-fold increase from baseline for pertussis toxin (and filamentous hemoglobin) and ≥ 10 mIU/mL for anti-HBs.

IPD SHARING:
Plan to Share IPD: No